CLINICAL TRIAL: NCT02850432
Title: The Evolution and Impact of Clinical and MRI Cardiac Biomarkers on Peripheral Arterial Disease in Patients With Long Term DM
Brief Title: Clinical and MRI Cardiac Biomarkers on Peripheral Arterial Disease in Patients With Long Term DM
Acronym: CMRPADDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsiang Juan, Primary investigator, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMRPG3F1311
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Magnetic resonance imaging; Extracellular volume matrix fraction; Peripheral artery disease; Blood-oxygen level dependent; Cardiac function
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Surgical Procedures, Operative; Conservative Treatment; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive treatment (Active Comparator): Endovascular therapy or surgery with medical therapy according to Trans-Atlantic Inter-Society Consensus II scoring system (TASC II)) as described in the main study protocol
  Interventions: Procedure: Invasive treatment
- Conservative treatment (Active Comparator): rehabilitation with medical therapy
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Procedure: Invasive treatment — Endovascular therapy or surgery with medical therapy according to Trans-Atlantic Inter-Society Consensus II scoring system (TASC II)) as described in the main study protocol
  Other Names: Surgery or endovascular treatment
  Arms: Invasive treatment
Other: Conservative treatment — rehabilitation with medical therapy
  Other Names: rehabilitation with medical therapy
  Arms: Conservative treatment

SUMMARY:
The aim of this study is to establish a clinically feasible simultaneous evaluation of heart and lower limb using MRI and to assess the combined benefit of clinical and cardiac MRI imaging markers in the evaluation of PAD and prediction of treatment outcome.

DETAILED DESCRIPTION:
We expect to enroll about 60 long-term DM patients (>10 years) from main study. Patient will receive evaluation of the perfusion in the lower limb by using blood oxygenation-level dependent (BOLD) sequence with measurement of the extracellular volume fraction (ECV) as an indicator of fibrosis severity in calf muscles. All patients will receive cardiac MRI (cardiac function, ischemia and fibrosis) and MR angiography (severity of PAD). The baseline studies will be completed within 2 years and 3 additional follow-up studies will be performed by the end of 4th year.

ELIGIBILITY:
The inclusion criteria include:

1. Able to understand and provide signed informed consent
2. DM history of 10 years and above
3. Willing to receive 3 MRI follow-up and serum hematocrit examinations within 2 years, if applicable
4. Willing to receive standard therapy such as surgery or medication
5. Age between 18-80 years old

The exclusion criteria include:

1. Pregnant or breast-feeding women
2. Allergic MRI contrast medium
3. Absolute contraindications to contrast MRI (e.g., metallic hazards, hemodynamic instability, pregnancy, known allergy to contrast medium).
4. Contraindicated to MRI study: cardiac pacemaker, cochlear implantation, metallic object within eyeball
5. Patients that refuse to, or has poor ability of understanding and comply study conditions, such as severe dementia or difficulty in mobility
6. Patients having dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-treatment improvement of peripheral artery disease | 2 years
  To determine the combined benefit of clinical and MRI imaging parameters (cardiac and lower extremities) in treatment response monitoring and treatment outcome prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Juan, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We have to see if this corresponds to the IRB regulation.

REFERENCES:
- [Derived] Lin YC, Fu TC, Lin G, Ng SH, Yeh CH, Ng SC, Chang TC, Juan YH. Using T1 mapping indices to evaluate muscle function and predict conservative treatment outcomes in diabetic patients with peripheral arterial disease. Eur Radiol. 2023 Jul;33(7):4927-4937. doi: 10.1007/s00330-023-09392-8. Epub 2023 Jan 18. PMID 36651955